CLINICAL TRIAL: NCT02033629
Title: Early Extubation After Cardiac Surgery: What Is the Appropriate Target Remifentanil Effect-Site Concentration?
Brief Title: Low Remifentanil Target Controlled Infusions for Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anesth-JAN14
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Surgery
Keywords: Anesthesia; remifentanil; propofol; target-controlled infusion; cardiac surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ce 1 ng/ml (Active Comparator): TCI Remifentanil Ce 1 ng/ml
  Interventions: Drug: Ce 1 ng/ml
- Ce 2 ng/ml (Active Comparator): TCI Remifentanil Ce 2 ng/ml
  Interventions: Drug: Ce 2 ng/ml
- Ce 3 ng/ml (Placebo Comparator): Remifentanil Ce 3 ng/ml
  Interventions: Drug: Ce 3 ng/ml

INTERVENTIONS:
Drug: Ce 1 ng/ml — TCI Remifentanil Ce 1 ng/ml
  Arms: Ce 1 ng/ml
Drug: Ce 2 ng/ml — TCI Remifentanil Ce 2 ng/ml
  Arms: Ce 2 ng/ml
Drug: Ce 3 ng/ml — TCI Remifentanil Ce 3 ng/ml
  Arms: Ce 3 ng/ml

SUMMARY:
The development of target effect-site controlled concentrations (TCI) of remifentanil have gained increasing acceptance during cardiac surgery as regarding the resulting of hemodynamic stability and early extubation. The use of low-dose opioid technique has been progressively used nowadays because of its ceiling effect to attenuate cardiovascular responses to noxious stimuli. We hypothesize that the use of low target remifentanil effect site concentrations may provide comparable shorter times to tracheal extubation and hemodynamic stability to the use of high remifentanil Ce during target-controlled propofol anesthesia for cardiac surgery.

DETAILED DESCRIPTION:
Reducing the time to tracheal extubation and hence the duration of postoperative mechanical ventilation could lessen postoperative complications, improve patients' outcome, shorten the intensive care unit (ICU) stay, and reduce the cost of treatment.

Although high-dose opioid cardiac anesthesia has been shown to provide hemodynamic stability and adequate depth of anesthesia in response to nociceptive stimulation, it may cause delayed recovery and lengthening of the durations for postoperative ventilation support and (ICU length of stay.

The pharmacokinetic-based drug infusion systems, target-controlled infusion (TCI), can rapidly and easily enables changes and maintenance of a constant blood concentration of intravenous anesthetic drugs. We demonstrated that, the use of a TCI of sufentanil at effect-site concentrations (Ce) from 0.2 to 0.3 ng/mL during TCI of propofol anesthesia for valve surgery shortened the times to clinical recovery and extubation.

Remifentanil, a short-acting opioid-receptor agonist with a context-sensitive half-time of 3 to 5 minutes allowing rapid emergence from anesthesia, even after an infusion of several hours. Compared with sufentanil (0.03 to 0.04 µg/kg/min), the use of remifentanil (0.5 to 1.0 µg/kg/min) during propofol anesthesia improved recovery of pulmonary function and shortened postoperative hospital length of stay after coronary artery bypass grafting (CABG).

Furthermore, a TCI of remifentanil at Ce of 1.5-5.0 ng/ml is more effective than a constant-rate infusion in the inhibition of the stress response and the maintenance of the cardiac autonomic nervous system balance during off-pump CABG. Similarly, the lowest remifentanil Ce used in another study of explicit and implicit memory during cardiac surgery under TCI propofol were 2 to 4 ng/ml.

Whereas, others used a wide range of remifentanil Ce from 2 to 10 ng/ml. However, the use of higher remifentanil Ce of 7 ng/ml (equivalent to 0.3 ng/kg/min) was associated with longer time to extubation than sufentanil Ce of 0.3 ng/ml (256 (92) vs. 161.9 (32.9) min, respectively).This precludes the favorable unique pharmacokinetic characteristics of remifentanil . Thus the use of low target controlled infusions of remifentanil could allow faster time to extubation and reduce the overall cost of the anesthetics.

We hypothesize that using low remifentanil target-controlled Ce during TCI of propofol anesthesia for cardiac surgery could decrease the time to tracheal extubation.

The subjects will be allocated randomly into the 3 groups by drawing sequentially numbered sealed opaque envelopes that each contained a software-generated randomization code.

The patients will be monitored by a pulse oximeter, 5-lead electrocardiograph (leads II and V5) with continuous ST-segment recording, radial mean arterial blood pressure (MAP) measurements, end-tidal carbon dioxide measurements, a central venous catheter or pulmonary artery catheter (according to the discretion of the attending anesthesiologist), and rectal and nasopharyngeal temperature measurements. Significant ischemic responses defined as reversible ST-segment changes from baseline, namely a ≥1-mV ST-segment depression or a ≥2-mV ST segment elevation that lasted for ≥1 minute. Response entropy (RE) and state entropy (SE) will be monitored by applying entropy electrodes (Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland) according to the manufacturer's recommendations.

An independent anesthesiologist who is not involved in collecting patient data will initiate the remifentanil Ce (the model of Minto et al) according to the patient's randomization code and is allowed to titrate the target propofol and remifentanil Ce and to administer vasoactive medications as needed. After preoxygenation, anesthesia induction by simultaneous target propofol and remifentanil infusions using the TCI system with syringe pumps (Injectomat TIVA Agilia, Fresenius Kabi, France).

The target propofol Ce (model of Schnider et al 13) will be initiated at 1.0 µg/mL and titrated stepwise by 0.5 µg/mL every 3 minutes until loss of consciousness and until an SE <50 and a difference <10 between RE and SE (RE-SE) will be achieved. Cisatracurium, 0.2 mg/kg, will be given to facilitate tracheal intubation, and the lungs will ventilated with a fraction of inspired oxygen of 0.5 to maintain normocapnia. The time from induction to intubation will be recorded.

Anesthesia will be maintained by changing the propofol Ce at increments of 0.5 µg/mL (range, 1-4.5 µg/mL) every 3 minutes as necessary to maintain an SE <50, RE-SE difference <10, and MAP and heart rate (HR) that are ≤20% of the baseline values. The remifentanil Ce will be increased by a maximum of 3 increments of 0.5 ng/mL when the SE is >50, the RE-SE difference is >10, and the MAP and HR are ≥20% of the baseline values despite a target propofol Ce >4.5 µg/mL. When the SE is <50 and the RE-SE difference is <10, the propofol Ce will be decreased gradually to ≥1 µg/mL, followed by gradual decreases in remifentanil Ce by 0.5 ng/mL, until the randomized Ce will be achieved. Based on our pilot study, the authors considered that using 0.5-ng/mL increments in remifentanil Ce would obtund the entropy and hemodynamic responses to noxious stimuli. The authors expected that 4 remifentanil Ce increments of 0.5 ng/mL would double the infusion rate in the Ce 1-ng/mL group to 2 ng/mL ([0.5 ng/mL x 4] + 1 ng/mL). The HR and MAP will kept within 20% of baseline values by achieving an adequate depth of anesthesia (SE <50 and RE-SE difference <10), optimum analgesia, and the administration of nitroglycerin, 0.05 mg, and esmolol, 20 mg. Cisatracurium, 1 to 3 µg/kg/min, was used to maintain surgical relaxation. All patients will receive tranexamic acid, 50 mg/kg.

Light anesthesia is defined as an episode with SE values >50 and/or MAP and HR values >20% above baseline that lasted for >3 consecutive minutes. The incidences of light anesthesia in response to intubation, skin incision, sternotomy, maximal sternal spread, and sternal wire placement will be recorded.

Hemodynamic control will be standardized according to the authors' protocol. Hypotension (defined as >20% decrease in mean baseline MAP) will be treated with boluses of fluids, phenylephrine 200 µg, ephedrine 5 mg, or epinephrine, 5 µg, as needed. Hypertension (defined as >20% increase in mean baseline MAP) will be treated by deepening anesthesia and administering doses of nitroglycerin, 0.05 mg, or labetalol, 20 mg. Tachycardia (defined as >20% increase in mean baseline HR) will be treated with esmolol, 20 mg.

All operations will be performed by the same surgeons. Heparin, 300 IU/kg, will be given to achieve an activated coagulation time >480 seconds. A standardized hypothermic cardiopulmonary bypass (CPB) will be used. The target propofol Ce and remifentanil Ce will be continued throughout surgery and CPB without any further adjustments because of CPB per se. Before separation from CPB, all patients will be rewarmed to a rectal temperature of 36°C and dobutamine, epinephrine, norepinephrine, and nitroglycerin will be used as needed. Heparin will be neutralized with protamine sulfate.

The cisatracurium infusion will be discontinued and morphine 0.1 mg/kg will be administered intravenously after surgical homeostasis is achieved. The target remifentanil Ce and propofol Ce will be discontinued after skin closure.

The HR, MAP, and cardiac and systemic vascular resistance indices will be recorded before (baseline) and 15 minutes after endotracheal intubation, 15 minutes after skin incision, 15 minutes after sternotomy, and 15 and 45 minutes after discontinuing CPB. Patients will be transferred to the intensive care unit (ICU) in a ventilated state using the synchronized intermittent mandatory mode or the pressure support mode.

Postoperative analgesia will be provided by intravenous paracetamol, lornoxicam, and patient-controlled analgesia (PCA), morphine 1 mg, with a lockout interval of 8 minutes and a maximum 4-hourly limit of 30 mg.

Extubation criteria included alertness, a train-of-four ratio ≥0.9, spontaneous breathing with a tidal volume >5 mL/kg, respiratory rates >10 and <28 breaths/min, a maximum inspiratory pressure ≤-20 cm H2O, stable hemodynamics without high doses of inotropic support or severe arrhythmias, bleeding <100 mL/h, a core temperature >35.5°C, a urine output >0.5 mL/ kg/h, an arterial carbon dioxide tension ≤45 mmHg, an arterial oxygen tension >100 mmHg, and a fraction of inspired oxygen <0.5. Blood samples will be drawn before CPB and 3, 12, 24, and 48 hours after CPB to measure cardiac troponin I levels.

Intraoperative explicit awareness will be assessed on the second postoperative day by asking the patients 3 simple questions in a standard interview: What was the last thing you remember happening before you went to sleep? What is the first thing you remember happening on waking? Did you dream or have any other experiences while you were asleep?

An independent investigator blinded to the study groups who is not involved in the patients' management will collect the patient data.

Sample size calculation:

A priori power analysis of the published data showed that the normally distributed mean time to tracheal extubation after remifentanil, 7 ng/mL, was 256 minutes (SD, 92 min). An a priori power analysis indicated that a sample size of 23 for each group was sufficiently large to detect 35% changes in the time to extubation after the administration of remifentanil Ce, 7 ng/mL, with a type-I error of 0.017 (0.05/3 possible comparisons) and a power of 90%. This sample size was increased by 10% to compensate for patients dropping out during the study.

In view of our amending our protocol on 2015 to compare the low remifentanil Ce 1, 2, and 3 ng/ml rather than the earlier considered 3 higher concentrations (2, 5, and 7 ng/ml) because of the noted significant haemodynamic compromise that required high use of inotropes/vasopressors, this earlier considered sample size calculation can not be valid anymore. Thus we recruited cases in a pilot study.

A pilot study showed that the normally distributed mean time to tracheal extubation after remifentanil, 3 ng/mL, was 39 minutes (SD, 14.92 min). An a priori power analysis indicated that a sample size of 21 for each group was sufficiently large to detect 15 min difference in the time to extubation after the administration of remifentanil Ce, 3 ng/mL, with a type-I error of 0.017 (0.05/3 possible comparisons) and a power of 90%. This sample size was increased by 10% to account for patients dropping out during the study.

Statistical Analysis

The data will be tested for normality using the Kolmogorov-Smirnov test. Repeated-measures analysis of variance will be used to analyze serial changes in the patient data at different times. The Fisher exact test will be used for categorical data. Repeated measures analysis of variance (ANOVA) will be used for continuous parametric variables and the differences will be corrected by the post hoc Bonferroni test. The Kruskal-Wallis test will be performed for intergroup comparisons for nonparametric values and post hoc pairwise comparisons were performed using the Wilcoxon rank-sum t test. The data will expressed as means (SD), number (percentage), or median [range]. A p value <0.05 is considered to represent statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* American Society of Anesthesiologists class III and IV
* eligible for early extubation

Exclusion Criteria:

* uncontrolled hypertension
* ischemic heart disease
* left ventricular ejection fraction ≤45%
* mean pulmonary artery pressure ≥50 mm Hg
* critical aortic stenosis
* pulmonary diseases
* hepatic diseases
* renal diseases
* neuromuscular diseases
* neuropsychiatric diseases
* endocrine diseases
* body mass index ≥40 kg/m2
* pregnancy
* use of antipsychotics
* use of alcohol
* drug abuse
* repeat surgery
* emergency surgery
* those requiring preoperative circulatory support
* those whose electrocardiographic characteristics would interfere with ST-segment monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-05; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
time to tracheal extubation | for 4 hours after surgery
  the times from skin closure to v

SECONDARY OUTCOMES:
times to spontaneous eye opening | for 5 hours during surgery
  times from skin closure to spontaneous eye opening
times from skin closure to return of spontaneous breathing | for 4 hours after surgery
  times from skin closure to return of spontaneous breathing (defined as a respiratory rate >12 breaths/min and an arterial oxygen saturation >95%);
the number of changes in propofol and remifentanil target infusions | for 6 hours during surgery
  the number of changes in propofol Ce and remifentanil Ce
Number of patients who will need changes in remifentanil effect site concentrations | For 6 hours during surgery
  the number of patients who will need changes in remifentanil Ce
rescue doses of medications | for 6 hours during surgery
  rescue doses of nitroglycerin, esmolol, phenylephrine, and ephedrine
incidences of light anesthesia | For 6 hours during surgery
  incidences of light anesthesia and awareness
Cost of Medications | for 6 hour during surgery
  Cost of Medications

CONTACTS AND LOCATIONS:
Locations (1):
- Dammam University, Khobar, Eastern Province, Saudi Arabia